CLINICAL TRIAL: NCT00917956
Title: A Pilot Trial of Lithium in Inclusion Body Myositis (IBM)
Brief Title: Lithium in Inclusion Body Myositis (IBM)
Acronym: Li-IBM
Status: Completed | Type: Observational
Sponsor: Phoenix Neurological Associates, LTD (Other)
Responsible Party: David Saperstein, MD, Phoenix Neurological Associates, LTD
Other Study IDs: WIRB #: 20071696; Study Number 1093885
Record Dates: First submitted 2009-06-08; First posted 2009-06-11 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: Inclusion Body Myositis
Keywords: Lithium; IBM; InclusionIBM; Myositis
MeSH Terms: conditions — Myositis, Inclusion Body; Myositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Muscle Biopsies will be taken at baseline and at the end of 6 months. Tissue will be frozen then sent out for anaylsis.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
IBM is the most common acquired muscle disease occurring over the age of 50. The underlying cause remains unknown and there is currently no effective treatment. Pathological studies have revealed abnormal collections of proteins in the muscle cells from patients with IBM. These include proteins called phosphorylated tau (p-tau). A similar process appears to occur in Alzheimer disease, with accumulations of p-tau developing in brain cells. Lithium decreases the activity of the GSK, an enzyme that has a key role in the development of p-tau. Lithium and other GSK inhibitors have been shown to decrease the accumulation of p-tau in nerve cells in animal models of Alzheimer disease. The proposed research is a pilot study to see if lithium might be an effective treatment for IBM

DETAILED DESCRIPTION:
Trial Status Open for Enrollment

What is the Purpose of this Study? There is currently no effective treatment for IBM and its pathogenesis remains uncertain. This study is designed to test the hypothesis that treatment of patients with IBM with Lithium can improve muscle strength and reduce the markers of disease activity believed to be important in the disease pathogenesis.

Who is Eligible to Participate? Patients diagnosed with Inclusion Body Myositis above the age of 30 who have adequate muscle function for quantitative muscle testing and who have a FVC >50%. Patients who have uncontrolled diabetes, renal insufficiency, congestive heart failure, cancer, hypothyroidism, current use of immunosuppressive medication, currently on warfarin or any known bleeding disorder are excluded.

What is involved in this Study? This is an open label trial looking at the effects of Li on muscle strength. Procedures consist of a baseline muscle biopsy, blood work, and other screening procedures. After the muscle biopsy patients are started on Li at 300mg/d. Lithium doses are dependent on tolerability and target lithium levels. Monthly visits consist of EKGs, Li level labs, questionnaires, and muscle strength testing. At month 6, patients will receive another muscle biopsy. The muscle biopsies are performed to analyze p-tau levels in the muscle.

How long is the Study? It is approximately 6 months long; however patients have the option to stay on the study for an additional 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >30
* Meet diagnostic criteria for definite IBM
* Muscle function adequate for quantitative muscle testing
* Able to give informed consent
* Women of child bearing potential must have a negative pregnancy test

Exclusion Criteria:

* Presence of uncontrolled diabetes, hypothyroidism, chronic infection, chronic renal insufficiency, congestive heart failure, cancer, or other chronic serious medical conditions
* Significant arrhythmias or conduction defect abnormalities on ECG
* Pregnant or lactating
* Coexistence of other neuromuscular or neurological diseases that would interfere with assessment
* Known bleeding disorder
* On Warfarin
* Contraindications to muscle biopsy: allergy to local anesthetic, skin infection, known bleeding disorder

Ages: 30 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who fit criteria diagnosed with IBM
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David D Saperstein, MD, Principal Investigator — Phoenix Neurological Associates, LTD
Locations (1):
- Phoenix Neurological Associates, LTD, Phoenix, Arizona, United States